CLINICAL TRIAL: NCT01569334
Title: Identification of Non Invasive Biomarkers of Immune Endothelial Injury and Repair Associated With Cardiac Allograft Vasculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-A01145-34; 2010 18 (Other: AP HM)
Record Dates: First submitted 2011-02-14; First posted 2012-04-03 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: identify early non invasive markers that index the endothelial lesion/ regeneration potential in association with CAV in heart transplanted recipients (HTR)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HTC with Cardiac allograft vasculopathy (Other): HTC:heart transplanted recipients
  Interventions: Biological: blood samples
- HTR without Cardiac allograft vasculopathy (Other)
  Interventions: Biological: blood samples
- untransplanted (Other)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples

SUMMARY:
Heart transplantation is the best option for patients with end-stage heart failure. Cardiac allograft vasculopathy (CAV) is the leading cause of death following cardiac transplantation and is not managed by current therapies. Its pathogenesis traduces in an accelerated form of coronary artery disease (CAD) with similarities to atherosclerosis but also particular features of endothelial dysfunction associated to the alloimmune conflict and humoral responses toward the graft. Intravascular ultrasound (IVUS) is the validated invasive method for late CAV diagnosis, but occurs lesions are established. Identification of reliable non-invasive early endothelial injury biomarkers that reflect mechanisms of cardiac damage thus remain a major challenge to optimize therapeutic management of post transplant morbidity. Endothelial dysfunction is a central feature of both CAV and CAD and results from a desquilibrium in the balance of endothelial lesion and repair that is partly controlled by recipient immune system. Through their expression of receptors sensing antibodies (FcR CD16) and endothelial stress-induced signals (CX3CR1 fractalkine receptor and NKG2D MICA receptors), Natural Killer (NK) cells represent effector cells with unique potential to generate both humoral and innate immune injury of graft endothelium.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years at the time of the inclusion,
* Subject having benefited from a heart transplant more than 11 months ago in the service of cardiac surgery concerned whatever is the treatment to immunosuppresseur current
* Subject benefiting from a coronarography within the framework of their surveillance comment-Clerk's Office beyond 12 months
* Subject having given their consent
* Affiliated to the Social Security

  * HTC with Cardiac allograft vasculopathy:
* Subject with coronaropathies diagnosed by the coronarography

  * TC without Cardiac allograft vasculopathy:
* Subject without coronaropathies diagnosed by the coronarography

  * untransplanted
* Untreated Subject by immunosuppresseurs
* Subject without antécédaent of transfusion
* Subject without history of transplantations
* Subject with coronaropathies diagnosed by a coronarography

Exclusion Criteria:

* Presenting a contraindication to the coronarography
* Subject refusing to practise the examination of coronarography
* Subject reaches(affects) of a cancer other one than cutaneous
* Subject achieves of hepatic Incapacity (ALAT and\or ASAT > 3N)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Analysis of endothelial lesion-repair biomarkers | 24 MONTHS
  through phenotypic and quantitative analysis of circulating endothelial progenitors subsets and (repair potential)

SECONDARY OUTCOMES:
Analysis of anti endothelial NK innate immune responses parameters | 24 MONTTHS
  * Anti endothelial, anti HLA anti MIC antibody detection in recipient' serum by luminex and flow cytometry
  * Evaluation of soluble Fractalkine and MIC levels in serum through ELISA
  * Analysis of CX3CR1 and CD16 polymorphism and phenotypic NK cell surface expression
  * Assay of serum induced and natural NK cell cytotoxicity against coronary and endothelial cell targets

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Paul P, Picard C, Sampol E, Lyonnet L, Di Cristofaro J, Paul-Delvaux L, Lano G, Nicolino-Brunet C, Ravis E, Collart F, Dignat-George F, Dussol B, Sabatier F, Mouly-Bandini A. Genetic and Functional Profiling of CD16-Dependent Natural Killer Activation Identifies Patients at Higher Risk of Cardiac Allograft Vasculopathy. Circulation. 2018 Mar 6;137(10):1049-1059. doi: 10.1161/CIRCULATIONAHA.117.030435. Epub 2017 Nov 2. PMID 29097449